CLINICAL TRIAL: NCT02109107
Title: An Evaluation of the Effect of the Erchonia® Zerona 6 Headed Scanner (EZ6) Six-week Treatment Protocol on Circumference Reduction of the Waist, Hips, Thighs and Upper Abdomen Clinical Study Protocol
Brief Title: Study of Low Level Laser Light Therapy on Circumference Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_EZ6_BC_001
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2015-12

CONDITIONS: Circumference Reduction
Keywords: body contouring; body shaping; circumference reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia EZ6 Laser (Experimental): The Erchonia EZ6 Laser is a 6 headed scanner composed of 6 independent 17 milliWatts (mW), 635 nanometer (nm) red laser diodes mounted in scanner devices. It is a variable frequency, pulsed wave laser device.
  Interventions: Device: Erchonia EZ6 Laser

INTERVENTIONS:
Device: Erchonia EZ6 Laser — The Erchonia EZ6 is administered 6 times across 6 consecutive weeks, each administration seven days apart, each treatment lasting 60 minutes.
  Other Names: Erchonia® Zerona 6 Headed Scanner

SUMMARY:
The purpose of this study is to determine whether low level laser light therapy is effective in reducing circumference of the waist, hips, thighs and upper abdomen over a 6 week period.

DETAILED DESCRIPTION:
The American Society of Plastic Surgeons (ASPS) 2011 report states that the market for cosmetic procedures has shown significant growth over the past two years, with 13.8 million cosmetic plastic surgery procedures performed in the United States in 2011, up 5% since 2010. While surgical cosmetic procedures significantly increased from 2010 to 2011, the overall growth in cosmetic procedures is primarily driven by a substantial rise in minimally-invasive procedures, that increased 6%, with nearly 12.2 million cosmetic minimally-invasive procedures having been performed in 2011. This highlights the growing consumer demand for non- or minimally-invasive cosmetic procedures that do not involve surgical procedures such as liposuction and the associated risks, potential complications and lengthy and painful recovery processes.

Low level laser light therapy offers a simple, non-invasive, safe, effective and side-effect free alternative to achieving body circumference reduction.

Justification for the assertion of anticipated safety and effectiveness of application of the Erchonia® EZ6 Laser low level laser therapy for the reduction of body circumference is found through three Food and Drug Administration (FDA) clearances for Erchonia® Low Level Laser devices for body circumference reduction indications, as follows:

K123237 (532 nanometer (nm) green light diodes): Erchonia® Zerona™ 2.0 Laser: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of hips, waist, and thighs.

K121695 & K082609 (635 nm red light diodes): Erchonia® ML Scanner (MLS) & Erchonia® Zerona: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of hips, waist, and thighs.

K121690 & K120257 (635 nm red light diodes): Erchonia® MLS, Zerona: is indicated for use as a non-invasive dermatological aesthetic treatment as an adjunct for individuals intending to undergo liposuction procedures for the reduction of circumference of the upper arms.

Therefore, Erchonia low level lasers have been determined safe and effective by the FDA for application for body circumference reduction indications for multiple body areas. The intended application/indication of the EZ6 in this study is comparable to the above FDA-cleared indications, with the study intent being to evaluate the comparative efficacy of a six week, once weekly 60 minute treatment administration protocol employing 6 red light diodes to the established efficacy of the current two week, thrice weekly 40 minute treatment administration protocol with application of five red light diodes on reduction of hips, waist, thighs and upper abdomen circumference.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 25 kg/m² and 40 kg/m²
* Subject indicated for liposuction or use of liposuction techniques for the removal of localized deposits of adipose tissues that do not respond to diet and exercise for the hips, waist, thighs and upper abdomen. (As per the American Academy of Cosmetic Surgery's 2006 Guidelines for Liposuction Surgery developed by A joint Ad Hoc Committee of the American Society of Lipo-Suction Surgery (ASLSS) and the American Academy of Cosmetic Surgery (AACS))
* Willing and able to abstain from treatments other than the study procedure for body contouring/circumference reduction/weight loss during study participation
* Willing and able to maintain typical diet and exercise regimen during study participation

Exclusion Criteria:

* Body Mass Index (BMI) less than 25 kg/m² or greater than 40 kg/m²
* Known cardiovascular disease
* Cardiac surgeries such as bypass, heart transplant surgery, pacemakers
* Prior surgical intervention for body sculpting/weight loss
* Medical, physical, or other contraindications for body sculpting/weight loss
* Current use of medication known to affect weight levels/cause bloating or swelling and for which abstinence during study participation is not possible
* Any medical condition known to affect weight levels and/or cause bloating or swelling.
* Diagnosis of, and/or taking medication for, irritable bowel syndrome.
* Active infection, wound or other external trauma to the study treatment areas
* Known photosensitivity disorder
* Active cancer or currently receiving treatment for cancer
* Pregnant or planning pregnancy prior to study participation end
* Serious mental health illness such as dementia/schizophrenia; psychiatric hospitalization in past two years.
* Developmental disability or cognitive impairment that may preclude adequate comprehension of the consent form and/or ability to record the study measures
* Involvement in litigation/worker's compensation/disability benefits related to the study parameters
* Participation in clinical research in the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl R Thornfeldt, MD, Principal Investigator; Paul M Thaxton, MD, Principal Investigator
Locations (2):
- United States (2):
  - Advanced Gynecology Specialists of Augusta, LLC, Evans, Georgia
  - CT Dermatology PC, Fruitland, Idaho

REFERENCES:
- [Derived] Thornfeldt CR, Thaxton PM, Hornfeldt CS. A Six-week Low-level Laser Therapy Protocol is Effective for Reducing Waist, Hip, Thigh, and Upper Abdomen Circumference. J Clin Aesthet Dermatol. 2016 Jun;9(6):31-5. Epub 2016 Jun 1. PMID 27386049

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia® Zerona 6 Headed Scanner (EZ6) Laser: The Erchonia® Zerona 6 Headed Scanner (EZ6) Laser is a 6 headed scanner composed of 6 independent 17 milliWatts (mW), 635 nanometer (nm) red laser diodes mounted in scanner devices. It is a variable frequency, pulsed wave laser device.
  Erchonia EZ6 Laser: The Erchonia EZ6 is administered 6 times across 6 consecutive weeks, each administration seven days apart, each treatment lasting 60 minutes.
Period: Overall Study
Arm/Group | Erchonia® Zerona 6 Headed Scanner (EZ6) Laser
Started | 54
Completed | 52
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia EZ6 Laser
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.39 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in Combined Circumference Measurements
Description: Combined circumference measurement is calculated as the sum of the measurements for the individual body areas of the right and left thighs, hips, waist and upper abdomen. Change in combined circumference measurements is calculated as the difference in measurements from baseline to after completion of the 6-week procedure administration period. A negative (-) change indicates a reduction in combined circumference measurement across the evaluation period and is positive for study success. A positive (+) change indicates an increase in combined circumference measurements across the evaluation period and is negative for study success.
  A mean change for the study subject group of -3.0 inches or more in combined circumference measurements will be considered a clinically meaningful and statistically significant positive change indicative of study success.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Erchonia EZ6 Laser
Number analyzed (Participants) | 54
inches | -5.36 (1.85)
Statistical Analysis 1: Comparison: Erchonia EZ6 Laser; Test type: Superiority or Other; p < .0001, t-test, 2 sided; t=21.33; df=53

2. Secondary Outcome: Change in Body Weight
Description: Body weight was measured in pounds at each evaluation point. The change in body weight measured in pounds at 6 weeks post-procedure administration relative to baseline was calculated. An increase in body weight indicated that weight was gained across the study evaluation period while a decrease in body weight indicated that weight was lost across the study evaluation period.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: pounds
Arm/Group | Erchonia EZ6 Laser
Number analyzed (Participants) | 54
pounds | -1.40 (0.85)
Statistical Analysis 1: Comparison: Erchonia EZ6 Laser; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; t=2.95; df=53

3. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Body mass index (BMI) was measured in kilograms per meter squared (kg/m2) at each evaluation point. The change in BMI measured at 6 weeks post-procedure administration relative to baseline was calculated. An increase in BMI indicated that BMI increased across the study evaluation period which is negative for study success, while a decrease in BMI indicated that BMI decreased across the study evaluation period which is positive for study success.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Erchonia EZ6 Laser
Number analyzed (Participants) | 54
kg/m2 | -0.28 (0.11)
Statistical Analysis 1: Comparison: Erchonia EZ6 Laser; Test type: Superiority or Other; p < 0.005, t-test, 2 sided; t+3.34; df=53

4. Secondary Outcome: Subject Satisfaction With Study Outcome Rating
Description: At the end of the study procedure administration phase, the subject was asked to indicate how satisfied or dissatisfied they were with any change noticed in the appearance of the thighs, hips, waist and upper abdomen area after having received the procedures with the EZ6?", using the following five-point scale: Very Satisfied; Somewhat Satisfied; Neither Satisfied nor Dissatisfied; Not Very Satisfied; Not at All Satisfied
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Erchonia EZ6 Laser
Number analyzed (Participants) | 52
participants
  Very Satisfied | 28
  Somewhat Satisfied | 14
  Neither Satisfied Nor Dissatisfied | 4
  Not Very Satisfied | 3
  Not At All Satisfied | 3

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Erchonia EZ6 Laser
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No